CLINICAL TRIAL: NCT06644300
Title: A Phase I, Multicenter, Non-randomized, Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of BM230 in Patients With Advanced Solid Tumors
Brief Title: Study of BM230 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Biomissile Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BM230-01
Record Dates: First submitted 2024-10-10; First posted 2024-10-16 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monotherapy BM230 Dose Escalation (Experimental): Patients will be treated with BM230 subcutaneous (s.c.) injection once every 1 week (Q1W) for 3 weeks in the 1st cycle and thereafter once every 2 weeks (Q2W) with 4 weeks as a cycle.
  Interventions: Drug: BM230
- Monotherapy BM230 Safety/PK/PD Expansion (Experimental): Expansion cohorts of monotherapy BM230 in multiple dose levels after evaluation for safety in Monotherapy Dose Escalation arm. Additional pharmacokinetic (PK) and pharmacodynamic (PD) samples included in this arm.
  Interventions: Drug: BM230

INTERVENTIONS:
Drug: BM230 — SC injection
  Arms: Monotherapy BM230 Dose Escalation
Drug: BM230 — SC injection
  Arms: Monotherapy BM230 Safety/PK/PD Expansion

SUMMARY:
This study is a Phase I, multicenter, non-randomized, open-label, first-in-human study of BM230 conducted globally. The study will include two parts: a dose escalation part (Phase Ia) followed by a dose expansion part (Phase Ib). Phase Ia part will estimate the MTD/RED(s) in dose escalation cohorts of patients with advanced solid tumors (HER2-related solid tumors). The Phase Ib part will enroll 5 distinct cohorts of patients with advanced solid tumors related to HER2 under MTD/RED doses, to better define the safety profile of BM230 and evaluate the efficacy of BM230.

ELIGIBILITY:
Inclusion Criteria:

Common inclusion criteria (Phase Ia and Phase Ib) (Criteria 1 to 9)

Patients must satisfy all the following criteria to be included in the study:

1. Informed of the study before any study-specific procedures are undertaken and voluntarily sign their name and date on the informed consent form (ICF)
2. Males and Females≥18 years old（at the time consent is obtained）
3. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 or 2
4. Life expectancy of ≥ 3 months
5. Adequate organ and bone marrow function, defined as:

   * Bone marrow function: hemoglobin ≥ 90 g/L (have not received blood transfusion or erythropoietin treatment within 14 days before the first dose); absolute neutrophil count ≥ 1.5×109/L (have not received granulocyte colony-stimulating factor or granulocyte-macrophage colony-stimulating factor treatment within 14 days before the first dose); platelet count ≥ 100×109/L ((have not received platelet transfusion, thrombopoietin, or interleukin-11 treatment within 14 days before the first dose)
   * Coagulation function: activated partial thromboplastin time and international normalized ratio ≤ 1.5 × ULN
   * Liver function (based on the normal range in the sites): TBIL ≤ 1.5 × ULN if no demonstrable liver lesion(s) (primary or metastases), or ≤ 3 × ULN in the presence of liver lesion(s), or < 4 × ULN for patients with Gilbert's syndrome; ALT and AST ≤ 3 × ULN if no demonstrable liver lesion(s) (primary or metastases), or ≤ 5 × ULN in the presence of liver lesion(s)
   * Renal function (based on the normal range in the sites): creatinine clearance (CrCl) calculated by the Cockcroft-Gault formula ≥ 50 mL/min, or 24-h urine CrCl ≥ 50 mL/min
   * Cardiac function: LVEF ≥ 50%;
6. Female patients of childbearing potential must agree to use a highly effective form of contraception and not donate, or retrieve for their own use, ova from the time of screening and throughout the study period, and for at least 6 months after the last dose of study drug; a negative pregnancy test must be obtained within 7 days before the first dose. Male patients must agree to use a highly effective form of contraception and not freeze or donate sperm from the time of screening and throughout the study period, and for at least 6 months after the last dose of study drug
7. Able and willing to comply with protocol visits and procedures
8. Have HER2 expression (IHC 1+, 2+, or 3+) determined by immunohistochemistry, or HER2 amplification (NGS report indicating HER2 amplification) or (for NSCLC) HER2 exon 8, exon 19, or exon 20 mutations. For Australia, only the cancer types with HER2 expression, amplification or mutation assay covered by Australia Pharmaceutical Benefits Scheme, and/or the patients with known HER2 expression, amplification or mutation obtained by any other program, will be considered to be enrolled
9. Willing to provide archived or fresh tumor tissue samples. Patients who are unable to provide tumor samples or have insufficient samples may be eligible on a case-by-case basis after discussion with the sponsor

   Additional inclusion criteria for Phase Ia (Criteria 10 to 11)
10. Pathologically confirmed diagnosis of locally advanced or metastatic solid tumors (BC, GC, CRC, and NSCLC are preferable), for which prior standard treatment had proven to be ineffective or intolerable, or no standard treatment is available, or the patient refuses standard treatment
11. Have at least one measurable tumor target lesion according to RECIST version 1.1. Patients in the accelerated titration cohort are not required for the above mentioned measurable tumor target lesion

    Additional inclusion criteria for Phase 1b (Criteria 12 to 13)
12. For Cohort A: BC patients:

    * Have a pathologically documented advanced/unresectable or metastatic BC
    * Have disease progression on or after the last treatment or intolerance to the last treatment, or for which no standard treatment is available

    For Cohort B: GC patients:
    * Have a pathologically documented advanced/unresectable or metastatic gastric or gastroesophageal junction adenocarcinoma
    * Have disease progression on or after prior treatment with at least one line of PD-(L)1 inhibitors and/or chemotherapy under metastatic setting

    For Cohort C: CRC patients:
    * Have a pathologically documented advanced/unresectable or metastatic CRC
    * Have disease progression on or after the last treatment or intolerance to the last treatment, or for which no standard treatment is available

    For Cohort D: NSCLC patients:
    * Have a pathologically documented Stage IIIB, IIIC, or IV squamous or non-squamous NSCLC
    * Have disease progression on or after prior anti-PD-(L)1 treatment and platinum-based chemotherapy
    * Have disease progression on or after prior on all targeted therapy for patients with mutations eligible targeted therapy

    For Cohort E (basket cohort): patients with other HER2-related solid tumors, including but not limited to ovarian cancer, endometrial cancer, cervical cancer, cholangiocarcinoma, pancreatic cancer, bladder cancer, and prostate cancer:

    • Have a pathologically documented advanced/unresectable or metastatic tumorHave disease progression on or after the last treatment or intolerance to the last treatment, or for which no standard treatment is available
13. At least one evaluable tumor target lesion according to RECIST version 1.1

Exclusion Criteria:

Patients who meet any of the following criteria will NOT be included in the study:

Common exclusion criteria (Phase Ia and Ib) (Criteria 1 to 19)

1. Preexisting autoimmune disease (except for patients with vitiligo) needing treatment with systemic immunosuppressive therapy for more than 28 days within the last 3 years, or clinically relevant immuno-deficiency diseases (eg, agammaglobulinemia or congenital immunodeficiency)
2. Multiple primary malignancies within 3 years, except adequately resected non-melanoma skin cancer, curatively treated in situ disease, or other curatively treated solid tumors (including but not limited to adequately treated thyroid cancer, carcinoma in situ of the cervix, basal or squamous cell skin cancer, or ductal carcinoma in situ of the breast treated with curative surgery)
3. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or in the follow-up period of an interventional study
4. In-sufficient washout period of the prior anticancer treatment before the first dose of the investigational product, defined as follows:

   * Anti-neoplastic treatments such as chemotherapy, biological therapy, nd immunotherapy within 3 weeks before the first dose
   * Radiotherapy for tumors within 2 weeks before the first dose
   * Endocrine therapy for tumors within 2 weeks before the first dose
   * Chinese herbal medicine or traditional Chinese medicine for tumor indications within 2 weeks before the first dose
   * Other investigational drugs or treatments within 4 weeks before the first dose (fluorouracil and small-molecule targeted drugs should be within 2 weeks before the first use of the investigational drugs or within 5 half-lives of the drug, whichever is shorter)
5. Undergone major surgery (not including diagnostic surgery) within 4 weeks before the first dose or are expected to undergo major surgery during the study
6. Undergone stem cell transplant or organ transplant
7. Received systemic corticosteroids (defined as > 10 mg/day of prednisone or equivalent) or other immuno-suppressive therapy within 2 weeks before the first dose. The following are exceptions to this criterion:

   * Intranasal, inhaled, topical steroids, topical corticosteroids or local steroid injections (eg, intra-articular injections)
   * Systemic steroids at physiological doses as replacement therapy (eg, physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency)
   * Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication)
8. Received any live vaccines within 4 weeks before the first dose or intend to receive live vaccines during the study
9. A history of leptomeningeal carcinomatosis; or existence of unstable central nervous system (CNS) metastases. Stability is defined as having undergone surgical resection and/or radiation therapy for CNS metastases at least 28 days before the first dose, and meeting all of the following criteria after completion of treatment:

   * No neurological symptoms, or symptoms are stable and ≤ grade 1
   * No progression of treated lesions and no new lesions within 28 days before the first dose by enhanced CT or magnetic resonance imaging (MRI) scan
   * Mild or no brain oedema on imaging during screening, but not requiring systemic corticosteroids or anti-convulsant drugs
10. Uncontrolled or clinically significant cardiovascular diseases, including but not limited to:

    * History of symptomatic CHF (New York Heart Association [NYHA] class II-IV) or any arterial embolism events (eg, myocardial infarction, unstable angina, cerebrovascular accident, and transient ischaemic attack) within 6 months before the first dose
    * Uncontrolled hypertension, defined as systolic blood pressure (SBP) >160 mmHg and/or diastolic blood pressure (DBP) >100 mmHg after antihypertensive treatment
    * Serious cardiac arrhythmia requiring treatment
    * The QT interval corrected by the Fridericia formula (QTcF) is prolonged to > 470 ms
11. Active haemorrhage with significant clinical significance
12. Uncontrolled third-space fluid (eg, pleural effusions, ascites, pericardial effusions) that requires repeated drainage
13. Uncontrolled or unstable systemic diseases, including diabetes mellitus, hepatic cirrhosis, interstitial lung disease, and obstructive lung disease, by the investigator's discretion
14. Uncontrolled infection that requires systemic therapy within 1 week before the first dose
15. Active hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV), or syphilis infection. Active HBV is defined as hepatitis B core antibody (HBcAb) or hepatitis B surface antigen (HBsAg) positive, and HBV DNA level above ULN at the study site; active HCV is defined as positive hepatitis C antibody and HCV RNA level above ULN at the site; active HIV is defined as positive HIV antibody; active syphilis is defined as positive Treponema pallidum lab test. Nevertheless, well-controlled HIV patients (deemed by the investigator) could be considered for enrollment
16. Unresolved toxicities from previous anticancer therapy, defined as toxicities not yet resolved to NCI CTCAE Grade ≤1, baseline, or the level specified in the inclusion/exclusion criteria with the exception of alopecia (any grade), pigmentation (any grade), and peripheral neuropathy (Grade ≤2). Patients with irreversible toxicity (eg, hearing loss) that is reasonably not expected to be aggravated by the study drug can be enrolled after discussion with the sponsor
17. A history of severe hypersensitivity reactions to the drug substances, inactive ingredients in the drug product, or other mAbs
18. Women who are breastfeeding or pregnant as confirmed by pregnancy tests performed within 7 days before the first dose
19. Any illness, medical condition, organ system dysfunction, or social situation, including but not limited to mental illness or substance/alcohol abuse, deemed by the investigator to be likely to interfere with a patient's ability to sign informed consent, adversely affect the patient's ability to cooperate and participate in the study, or compromise the interpretation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
DLT | 21 days
  Dose limiting toxicity
AEs | up to 3 years
  Adverse events
MTD and/or RED | up to 3 years
  The maximum tolerated dose (MTD) and/or the recommended expansion dose

SECONDARY OUTCOMES:
AUC | up to 3 years
  area under the concentration-time curve
Cmax | up to 3 years
  maximum concentration
Ctrough | up to 3 years
  trough concentration
CL | up to 3 years
  clearance rate
Vd | up to 3 years
  volume of distribution
t1/2 | up to 3 years
  half-life time
ADA | up to 3 years
  Anti-drug antibody
ORR | up to 3 years
  Objective response rate assessed using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
DCR | up to 3 years
  Disease control rate (DCR) assessed using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
DoR | up to 3 years
  Duration of response (DoR) assessed using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
BOR | up to 3 years
  Best overall response (BOR) assessed using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
TTR | up to 3 years
  Time to response (TTR) assessed using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
PFS | up to 3 years
  Progression-free survival (PFS) assessed using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
OS | up to 3 years
  Overall survival (OS) assessed using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (3):
  - Icon Cancer Centre - South Brisbane, Brisbane, Queensland
  - Southern Oncology Clinical Research Unit, Adelaide, South Australia
  - Monash Health - Monash Medical Centre, Monash, Victoria
- China (3):
  - The first Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - Fudan Unversity Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang